CLINICAL TRIAL: NCT02616549
Title: A Randomized Study of a Comprehensive Yoga Intervention for Patients With Major Depressive Disorder With Incomplete Response to Antidepressants
Brief Title: Multicomponent Yoga Intervention for Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 820672
Record Dates: First submitted 2015-11-23; First posted 2015-11-30 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sudarshan Kriya Yoga (Experimental)
  Interventions: Behavioral: Sudarshan Kriya Yoga
- Waitlist Control (No Intervention)

INTERVENTIONS:
Behavioral: Sudarshan Kriya Yoga — A manual-based yoga program featuring a yoga-breathing meditation technique
  Arms: Sudarshan Kriya Yoga

SUMMARY:
The purpose of this study is to evaluate the efficacy of a multi-component yoga intervention featuring Sudarshan Kriya Yoga (SKY) as an adjunctive treatment for patients with Major Depressive Disorders with incomplete response to antidepressants.

DETAILED DESCRIPTION:
According to the World Health Organization, compared to two hundred health conditions, depression is ranked as the second leading cause of disability worldwide. The annual prevalence of Major Depressive Disorder (MDD) in the United States is estimated at 7% and the lifetime risk approximately 17%. Depression is associated with approximately 75% of all deaths by suicide, resulting in immense suffering for families and society at large. 83 billion dollars are spent per year on treatment and lost productivity related to the disorder. Current treatments for MDD have remission rates between 35-50%. Patients who respond to treatment, but do not experience clinical remission are at markedly increased risk for relapse. Approximately 50% of patients treated with two trials of antidepressant interventions do not achieve clinical remission. Consequently, novel evidence-based treatment modalities that can further treat this devastating disorder are needed. Mind-body interventions constitute a large and diverse group of practices that reduce both stress and inflammation and are increasingly being evaluated in the treatment of MDD The 2007 NHIS concluded that 16.6% of U.S. adults, representing 34.1 million Americans, used at least one mind-body intervention in the past year. Initial studies with different mind-body interventions have been shown to improve outcomes in MDD. A recent meta-analysis gave a Grade B for current evidence for the use of yoga as an intervention for MDD. Sudarshan Kriya Yoga (SKY) is a advanced yogic breathing intervention that has been reported to relieve symptoms of major depressive disorder and generalized anxiety disorder. In MDD, SKY can correct the P300 amplitude, decrease plasma cortisol levels and increase plasma prolactin levels. In a small-scale randomized controlled trial, 45 consenting inpatients meeting criteria for DSM-IV severe, melancholic depression were randomized to receive SKY, electroconvulsive therapy (ECT) or imipramine treatment for four weeks (Janakiramaiah et al. 2000). Consequently, the rigorous evaluation of a multicomponent yogic intervention featuring SKY as an adjunctive treatment for adults with MDD warrants further study.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Major Depressive Disorder
* Able to give informed consent
* Aged 18-67
* Currently in outpatient care for MDD
* On a stable antidepressant regimen for at least 2 months
* 17-item Hamilton Depression Score >14 at screening & baseline visit

Exclusion Criteria:

* Currently in crisis requiring inpatient treatment
* Bipolar Disorder, Psychotic Disorder, ADHD, Substance Use Disorder
* Pregnancy, Epilepsy
* Initiating psychotherapy or other yoga/meditation program

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
17-item Hamilton Depression Rating Scale | Baseline to 2 month

SECONDARY OUTCOMES:
Beck Depression Inventory | Baseline to 2 month
Beck Anxiety Inventory | Baseline to 2 month
Columbia Suicide Severity Rating Scale | Baseline, 1 month, 2 month

OTHER OUTCOMES:
Serum Inflammatory Markers | Baseline, 1 month, 2 month

CONTACTS AND LOCATIONS:
Locations (1):
- Mood & Anxiety Disorders Research and Treatment Program, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Sharma A, Barrett MS, Cucchiara AJ, Gooneratne NS, Thase ME. A Breathing-Based Meditation Intervention for Patients With Major Depressive Disorder Following Inadequate Response to Antidepressants: A Randomized Pilot Study. J Clin Psychiatry. 2017 Jan;78(1):e59-e63. doi: 10.4088/JCP.16m10819. PMID 27898207